CLINICAL TRIAL: NCT03986281
Title: A Pilot Study to Assess the Accuracy of Blood Pressure Assessment by the Omron HeartGuide Smartwatch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Marc Gillinov, MD, Principal Investigator, The Cleveland Clinic
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 19-319
Record Dates: First submitted 2019-06-12; First posted 2019-06-14 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Hypertension; Cardiac Disease; Surgery
Keywords: Wearable devices; Blood pressure; Arterial line; Hypertension; Post Operative; Cardiac Surgery
MeSH Terms: conditions — Hypertension; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omron HeartGuide Smartwatch (Active Comparator): Readings from the Omron HeartGuide Smartwatch
  Interventions: Other: Omron Wearable Device
- Arterial Line (Active Comparator): Readings from the arterial line
  Interventions: Other: Standard Arterial Line

INTERVENTIONS:
Other: Omron Wearable Device — Omron wearable device compared to arterial line readings
  Arms: Omron HeartGuide Smartwatch
Other: Standard Arterial Line — Omron wearable device compared to arterial line readings
  Arms: Arterial Line

SUMMARY:
The accuracy of devices like the recent FDA-clearance of the Omron HeartGuide™ Blood Pressure sensor in robust clinical settings remain in question and thus form the underpinning of this research study.

The objective of this pilot prospective study is to assess the accuracy of the Omron Blood Pressure sensor as compared to arterial line blood pressure monitoring.

DETAILED DESCRIPTION:
The purpose of this study is to assess the accuracy of the Omron HeartGuide™ Smartwatch in measuring blood pressure and heart rate as compared to standard post-operative blood pressure and heart rate monitoring with an arterial line and heart monitor.

Hypertension affects about 75 million Americans and is the leading cause of cardiovascular disease (heart attacks and strokes), resulting in about 1,000 deaths per day. Only 50% of patients have their blood pressure adequately managed thus necessitating a better solution. Current limitations to hypertension management in non-ICU or non-surgical settings include: 1) infrequent measurements, 2) inherent data variability, 3) white coat hypertension, 4) non-compliance, or 5) poor patient-provider follow-up. A majority of patients have their blood pressure measured only during clinic visits. A wearable blood pressure sensor that takes multiple measurements per day will allow for a new level of granularity among measurements. With more continuous measurements, patients and physicians can work together to identify the onset and progression of hypertension before it causes irreversible damage to the heart, kidneys, and brain.

During testing, each subject will wear the Omron HeartGuide™ Smartwatch. Both right and left wrist circumferences will be measured prior to placing the device. All patients will be on continuous telemetry according to standard clinical practice on the ICU. Each patient will be outfitted with the Omron HeartGuide™ Smartwatch (opposite extremity of the arterial line). An Omron BP reading will be obtained at the same time as the arterial line reading. Four readings in total will be obtained for each patient. All four readings may occur on the same day or may be occur over several days.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Post-operative cardiac surgery patients on the ICU floors at the Cleveland Clinic Main Campus
* Wrist size range ranging from 16 cm to 19 cm

Exclusion Criteria:

* Wrist size range smaller than 16 cm or larger than 19 cm
* Use of a radial artery graft for coronary artery bypass grafting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Accuracy of the Omron blood pressure sensor | 24 hours
  Omron device accuracy as compared to arterial line BP readings

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gillinov, M. D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuwabara M, Harada K, Hishiki Y, Kario K. Validation of two watch-type wearable blood pressure monitors according to the ANSI/AAMI/ISO81060-2:2013 guidelines: Omron HEM-6410T-ZM and HEM-6410T-ZL. J Clin Hypertens (Greenwich). 2019 Jun;21(6):853-858. doi: 10.1111/jch.13499. Epub 2019 Feb 25. PMID 30803128